CLINICAL TRIAL: NCT04693728
Title: Adaptive Strategies for Resilient Intrinsic Self-Regulation in Extremes (RISE): A Controlled Clinical Trial as an Intervention for Chronic Pain From a Homeostatic Perspective
Brief Title: Adaptive Strategies for Resilient Intrinsic Self-Regulation in Extremes (RISE)
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phoenix VA Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Aram Mardian, Senior Research Scientist, Phoenix VA Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1054
Record Dates: First submitted 2020-12-23; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention (Active Comparator): The study intervention arm was a behavioral treatment that consisted of training resilient intrinsic self-regulation strategies to help alleviate chronic pain.
  Interventions: Behavioral: Resilient Intrinsic Self-Regulation Strategies in Extremes
- Wait-list with no treatment (No Intervention): The control comparison arm consisted of a wait-list condition in which participants received no treatment during a time interval comparable to the intervention arm.

INTERVENTIONS:
Behavioral: Resilient Intrinsic Self-Regulation Strategies in Extremes — The manualized intervention covered resilience strategies organized into four modules: (1) engagement, (2) social relatedness, (3) transformation of pain and (4) building a good life. The modules were delivered in 8 weekly sessions of 90 minutes each.
  Other Names: Active Intervention arm
  Arms: Behavioral Intervention

SUMMARY:
The purpose of this study is to assess the efficacy of a resilience intervention in Veterans with chronic pain compared to wait list control.

DETAILED DESCRIPTION:
After being consented and screened for eligibility, participants completed baseline assessments and then were randomized to either the study intervention or wait list control. Participants who were randomized to the study intervention completed post testing assessment measures within two weeks of the final treatment. Participants who were randomized to waitlist conditions completed post testing assessment measures within 2 weeks of the end of the waitlist condition and then subsequently received the study intervention.

ELIGIBILITY:
Inclusion Criteria:

1.18-80 years of age 2. United States Veterans from the conflicts of OEF/OIF to Vietnam era 3. Self-identified chronic pain or chart diagnosis of chronic pain

Exclusion Criteria:

1. Active suicidality of suicidal intent requiring a greater than outpatient level of care (Columbia Suicidality Rating Scale screen, C-SSRS)
2. Active alcohol abuse (Alcohol Use Disorder Identification Test, AUDIT-C)
3. Active psychosis (Psychosis Screener)
4. Current severe disabling illness
5. Inability to participate in a small group interactive setting
6. Inability to meet attendance requirement
7. Neurocognitive conditions other than TBI (e.g. dementia, Parkinsons, stroke)
8. Concurrently receiving Exposure Therapy, Cognitive Behavior Therapy, Acceptance and Commitment Therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-08-13 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
RAND 36-item Health Survey (SF-36) - Mental Health and Physical Health subscales | 2 weeks
  assessment of positive emotional health
PTSD Check List-5 | 2 weeks
  assessment of PTSD symptoms
Patient Health Questionnaire, Depression Scale (PHQ-9) | 2 weeks
  assessment of depression symptoms
Generalized Anxiety Disorder (GAD-7) | 2 weeks
  assessment of anxiety symptoms
Pain Catastrophizing Scale | 2 weeks
  assessment of pain catastrophizing symptoms
Physical Symptoms Scale (PHQ-15) | 2 weeks
  assessment of physical symptoms
Insomnia Severity Index | 2 weeks
  assessment of insomnia symptoms
West Haven-Yale Multidimensional Pain Inventory (WYMPI) | 2 weeks
  multidimensional assessment of pain
Pain Outcomes Questionnaire (POQ) | 2 weeks
  multidimensional assessment of pain
Neuropsychological Assessment Battery (NAB) - Word Generation subtest | 2 weeks
  neuropsychological assessment of executive functions
Delis-Kaplan Executive Function System (D-KEFS) - Category Fluency, Category Switching, and Color-Word Switching subtests | 2 weeks
  neuropsychological assessement
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | 2 weeks
  neuropsychological assessment of working memory, episodic memory, and complex attention

CONTACTS AND LOCATIONS:
Overall Officials: Martha Kent, PhD, Principal Investigator — Phoenix VAHCS
Locations (1):
- Phoenix VA Health Care System, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kent M, Mardian AS, Regalado-Hustead ML, Gress-Smith JL, Ciciolla L, Kim JL, Scott BA. Adaptive Homeostatic Strategies of Resilient Intrinsic Self-Regulation in Extremes (RISE): A Randomized Controlled Trial of a Novel Behavioral Treatment for Chronic Pain. Front Psychol. 2021 Apr 12;12:613341. doi: 10.3389/fpsyg.2021.613341. eCollection 2021. PMID 33912102